CLINICAL TRIAL: NCT07354126
Title: Comparative Efficacy of Flunarizine and Propanolol in Pediatric Migraine Using the PedMIDAS Measuring Tool.
Brief Title: Comparative Efficacy of Flunarizine and Propanolol in Pediatric Migraine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dr-Ishfaq-Lhr
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Flunarizine; Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flunarizine group (Experimental): Patients will be receiving flunarizine beginning with 5 mg at bedtime and increasing it to 10 mg at bedtime after 1 month, over a 3-month treatment period.
  Interventions: Drug: Flunarizine
- Propranolol group (Experimental): Patients will be given propranolol beginning with 10 mg/24 hours and increasing at the rate of 10 mg/week to the maximum of 60 mg/24 hours over a 3-month treatment period.
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Flunarizine — Patients will be receiving flunarizine beginning with 5 mg at bedtime and increasing it to 10 mg at bedtime after 1 month, over a 3-month treatment period.
  Arms: Flunarizine group
Drug: Propranolol — Patient will be given propranolol beginning with 10 mg/24 hours and increase at the rate of 10 mg/week to the maximum of 60 mg/24 hour, over a 3-month treatment period.
  Arms: Propranolol group

SUMMARY:
Flunarizine and propranolol have demonstrated efficacy in reducing migraine frequency across age groups, though evidence in pediatric populations remains limited and inconsistent. Therefore, the current study has been planned to evaluate and compare the effectiveness of flunarizine and propranolol in reducing migraine frequency in children aged 8-15 using the Pediatric Migraine Disability Assessment Scale (PedMIDAS) score.

DETAILED DESCRIPTION:
Despite the clinical use of flunarizine and propranolol, direct comparisons between these two drugs in children are scarce. This study aims to bridge that gap by evaluating their relative effectiveness and safety as prophylactic treatments for pediatric migraine, addressing a critical unmet need in current research. Considering the routine use of both drugs in clinical practice, the findings would help clinicians to choose the more convenient drug between flunarizine and propranolol as preventive therapy for migraine in their local settings.

ELIGIBILITY:
Inclusion Criteria:

* Children of any gender
* Aged 8-15 years
* Diagnosed with migraine (with/without aura) per International Classification of Headache Disorders, 3rd Edition (ICHD-3) criteria
* A history of ≥4 migraine attacks/month for the preceding 3 months
* With a PedMIDAS score ≥11 (moderate-to-severe impact)

Exclusion Criteria:

* Children with secondary headache disorders (e.g., due to infections, trauma, structural brain lesions)
* Known hypersensitivity or contraindications to flunarizine or propranolol
* Presence of cardiovascular disorders (e.g., bradycardia, heart block, hypotension, asthma)
* Non-compliance or inability to attend regular follow-ups
* Participation in another clinical trial within the last 3 months

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Reduction in migraine disability | 3 months
  Any reduction in migraine disability score measured by PedMIDAS will be labeled as reduction (efficacy).

CONTACTS AND LOCATIONS:
Overall Officials: Ishafaq Ahmed, FCPS, Principal Investigator — The Children's Hospital Lahore; Muhammad Zia-ur-Rehman, FCPS, Study Director — The Children's Hospital Lahore
Locations (1):
- The Children's Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.